CLINICAL TRIAL: NCT03526757
Title: The Effects of Pilates Standing Exercises on Walking Mobility and Postural Balance in Sedentary Older Adults: a Randomized Clinical Trial
Brief Title: Effects of Pilates Standing Exercises on Walking Mobility and Postural Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 8185
Record Dates: First submitted 2018-04-26; First posted 2018-05-16 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2019-07

CONDITIONS: Aging; Mobility Limitation; Postural Balance
Keywords: Postural balance; Pilates method; Elderly
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: The subjects will be allocated to one of two groups: intervention protocol (high volume of standing Pilates exercises) or control protocol (standard sequence of Pilates exercises).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are masked for subject allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing Pilates protocol (Experimental): Subjects will be submitted to a bi-weekly, 50-minute session of Pilates exercises focusing on orthostatic position, for twelve weeks. The following equipment will be used: The Cadillac, Reformer and Chair, emphasizing balance training in the orthostatic position.
  Interventions: Other: Standing Pilates protocol
- Standard Pilates protocol (Active Comparator): Subjects will be submitted to a bi-weekly, 50-minute session of the standard sequence of Pilates exercises (traditional sequence of the contemporary / classical method) for twelve weeks. The exercises will be performed using the same equipment used in the intervention group, but following the dorsal decubitus, sedestation and orthostasis, in a time-balanced distribution in each session.
  Interventions: Other: Standard Pilates protocol

INTERVENTIONS:
Other: Standing Pilates protocol — Subjects will be submitted to a bi-weekly, 50-minute session of Pilates exercises focusing on orthostatic position, for twelve weeks. The following equipment will be used: The Cadillac, Reformer and Chair, emphasizing balance training in the orthostatic position.
  Other Names: Pilates exercises in orthostatic position
  Arms: Standing Pilates protocol
Other: Standard Pilates protocol — Subjects will be submitted to a bi-weekly, 50-minute session of the standard sequence of Pilates exercises (traditional sequence of the contemporary / classical method) for twelve weeks. The exercises will be performed using the same equipment used in the intervention group, but following the dorsal decubitus, sedestation and orthostasis, in a time-balanced distribution in each session.
  Other Names: Standard Pilates exercises
  Arms: Standard Pilates protocol

SUMMARY:
Importance: Aging is characterized by numerous molecular, physiological, functional, motor and psychological changes, such as loss of postural balance and reduced muscle mass/strength. Such modifications often lead to reduced physical-functional capacity in the elderly and increased risk of falls. Currently, physical exercise is widely used to improve physical performance and reduce, at least in part, postural instabilities and the risk of falls. In this context, the Pilates method may be a good strategy to improve body balance, muscle strength and, potentially, the perception of quality of life in this population, depending how the exercises are performed. This study seeks to assess whether practicing Pilates exercises in orthostatic position results in differential effects on walking mobility and postural balance in healthy elderly women when compared to the standard sequence in the Pilates method, which involves less time performing exercise in the orthostatic position. The study hypothesis is that a higher relative volume of Pilates exercises performed in the orthostatic position can promote greater benefits in terms of walking mobility and postural balance compared to the standard Pilates protocol in the elderly.

DETAILED DESCRIPTION:
Importance: Aging is characterized by numerous molecular, physiological, functional, motor and psychological changes, such as loss of postural balance and reduced muscle mass/strength. Such modifications often lead to reduced physical-functional capacity in the elderly and increased risk of falls. Currently, physical exercise is widely used to improve physical performance and reduce, at least in part, postural instabilities and the risk of falls. In this context, the Pilates method may be a good strategy to improve body balance, muscle strength and, potentially, the perception of quality of life in this population, depending how the exercises are performed.

Objective: To evaluate whether practicing Pilates exercises in orthostatic position results in differential effects on walking mobility and postural balance in healthy elderly women when compared to the standard sequence in the Pilates method, which involves less time performing exercise in the orthostatic position.

Design, Methods and Participants: Clinical, single blind controlled and randomized trial. 36 previously sedentary elderly women will be included in the study and sign a Free and Informed Consent Term (TCLE). The Pilates protocols will be administered over 12 weeks on a bi-weekly scheme, and each session will last approximately 50 minutes. The subjects who agree to participate will be evaluated at baseline and immediately post-intervention.

Intervention: Subjects will be randomized to participate in the experimental group (Pilates exercises with emphasis on orthostatic posture) or control group (Pilates exercises practiced following traditional sequence of postures).

Main Outcomes and Measurements: The main outcome of the study will be walking mobility and postural balance, assessed using the Timed Up and Go test (single "motor" and dual task "cognitive-motor" tests), BERG Balance Scale, Functional Reach Test, and ABC Balance Confidence Scale).

Expected results: The experimental group is expected to perform better in terms of walking mobility and body balance, since hypothetically, a higher relative volume of orthostatic exercises would be more adequate for training anticipatory postural adjustments when compared to the traditional Pilates postural sequence.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary for at least 6 months
* To be available for one hour, twice a week, on two different working days to perform the proposed exercises.
* To show preserved cognitive function, according to the mini-mental state examination criteria;
* Be able to come and go on their own to the training location (Physiotherapy Laboratory at PUCRS).

Exclusion Criteria:

* Clinical contraindications for performing physical exercises;
* To show severe heart, orthopedic, neurological or other diseases/conditions that may affect the outcome measures;
* Practicing physical exercises outside the study protocol;
* Absence of independent gait.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study seeks to investigate elderly women, since they show higher risk of falling.
Enrollment: 36 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Walking mobility (Timed Up and Go Test) | Post-intervention (change after 12 weeks of training)
  Walking mobility will be assessed using the Timed Up and Go tests (single and dual task - cognitive/motor). It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require.

SECONDARY OUTCOMES:
Postural balance - Functional Reach Test | Post-intervention (change after 12 weeks of training)
  Postural balance will be assessed using the Functional Reach Test. The FRT is a quick single-task dynamic test defined as the maximal distance one can reach forward beyond arm's length, while maintaining a fixed base of support in the standing position.
Postural balance - BERG Balance scale | Post-intervention (change after 12 weeks of training)
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Activities-specific Balance Confidence (ABC) Scale. | Post-intervention (change after 12 weeks of training)
  For each assessed activity, the subjects indicate their level of confidence in doing the activity without losing your balance or becoming unsteady from choosing one of the percentage points on the scale from 0% to 100%. If subjects do not currently do the activity in question, they should imagine how confident they would be if had to do the activity. If they normally use a walking aid to do the activity or hold onto someone, subjects should rate their confidence as if they were using these supports.
Quality of life (36-Item Short Form Health Survey - SF-36) | Post-intervention (change after 12 weeks of training)
  Quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). The SF-36 consists of eight scaled scores (vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; and mental health.), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

OTHER OUTCOMES:
Physical Activity Levels | Baseline
  Physical Activity Levels will be assessed using the International Physical Activity Questionnaire (IPAQ). The International Physical Activity Questionnaire (IPAQ) estimates the weekly energy expenditure for physical activities (PA). This instrument was validated for use with Brazilian older adults. The report of the IPAQ adapted for older adults should be delivered in minutes per week.
Cognition screening | Baseline
  Cognitive decline will be screened using the Mini Mental State Examination (MMSE). The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age. That is, a maximal score of 30 points can never rule out dementia. Low to very low scores correlate closely with the presence of dementia, although other mental disorders can also lead to abnormal findings on MMSE testing.
Depression screening | Baseline
  Depression will be screened using the Geriatric Depression Scale (GDS). The scale consists of 30 yes/no questions. Each question is scored as either 0 or 1 points. The following general cutoff may be used to qualify the severity: 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".

CONTACTS AND LOCATIONS:
Overall Officials: Régis G Mestriner, PhD, Study Chair — Pontifícia Universidade Católica do Rio Grande do Sul
Locations (1):
- Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We will make all efforts to publish and make individual participant data (IPD) available, according to the requirements of the scientific journal that accepts this research.

REFERENCES:
- [Background] Bird ML, Hill KD, Fell JW. A randomized controlled study investigating static and dynamic balance in older adults after training with Pilates. Arch Phys Med Rehabil. 2012 Jan;93(1):43-9. doi: 10.1016/j.apmr.2011.08.005. Epub 2011 Oct 5. PMID 21975148
- [Background] Walowska J, Bolach B, Bolach E. The influence of Pilates exercises on body balance in the standing position of hearing impaired people. Disabil Rehabil. 2018 Dec;40(25):3061-3069. doi: 10.1080/09638288.2017.1370731. Epub 2017 Nov 13. PMID 29132250
- [Background] Bueno de Souza RO, Marcon LF, Arruda ASF, Pontes Junior FL, Melo RC. Effects of Mat Pilates on Physical Functional Performance of Older Adults: A Meta-analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2018 Jun;97(6):414-425. doi: 10.1097/PHM.0000000000000883. PMID 29283899
- [Background] Oliveira LC, Oliveira RG, Pires-Oliveira DAA. Pilates increases the isokinetic muscular strength of the knee extensors and flexors in elderly women. J Bodyw Mov Ther. 2017 Oct;21(4):815-822. doi: 10.1016/j.jbmt.2017.01.006. Epub 2017 Jan 8. PMID 29037633
- [Background] Bertoli J, Biduski GM, de la Rocha Freitas C. Six weeks of Mat Pilates training are enough to improve functional capacity in elderly women. J Bodyw Mov Ther. 2017 Oct;21(4):1003-1008. doi: 10.1016/j.jbmt.2016.12.001. Epub 2016 Dec 3. PMID 29037615
- [Background] Teixeira de Carvalho F, de Andrade Mesquita LS, Pereira R, Neto OP, Amaro Zangaro R. Pilates and Proprioceptive Neuromuscular Facilitation Methods Induce Similar Strength Gains but Different Neuromuscular Adaptations in Elderly Women. Exp Aging Res. 2017 Oct-Dec;43(5):440-452. doi: 10.1080/0361073X.2017.1369624. Epub 2017 Sep 26. PMID 28949820
- [Background] Vieira ND, Testa D, Ruas PC, Salvini TF, Catai AM, de Melo RC. The effects of 12 weeks Pilates-inspired exercise training on functional performance in older women: A randomized clinical trial. J Bodyw Mov Ther. 2017 Apr;21(2):251-258. doi: 10.1016/j.jbmt.2016.06.010. Epub 2016 Jun 21. PMID 28532866
- [Background] Greblo Jurakic Z, Krizanic V, Sarabon N, Markovic G. Effects of feedback-based balance and core resistance training vs. Pilates training on cognitive functions in older women with mild cognitive impairment: a pilot randomized controlled trial. Aging Clin Exp Res. 2017 Dec;29(6):1295-1298. doi: 10.1007/s40520-017-0740-9. Epub 2017 Mar 1. PMID 28251569